CLINICAL TRIAL: NCT05858216
Title: First-generation OTC Antihistamine Use and Voice Function: A Preliminary Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Mary J. Sandage, Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-175
Record Dates: First submitted 2023-04-26; First posted 2023-05-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Voice Disorder Due to Iatrogenic Factor
MeSH Terms: interventions — Chlorpheniramine

STUDY DESIGN:
Intervention Model Description: Within participant repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chlor-Trimeton (Other): Package recommended dose of over the counter Chlor-Trimeton will be administered to assess voice function before and 3 hours after taking it.
  Interventions: Drug: Chlor-Trimeton.

INTERVENTIONS:
Drug: Chlor-Trimeton. — Package dose of Chlor-Trimeton will be administered

SUMMARY:
The goal of this clinical trial is to learn about voice function before and 3 hours after administration of first generation over-the-counter antihistamine in individuals who have been medically diagnosed with allergies and routinely take over-the-counter (OTC) antihistamines for allergy symptoms. The main questions are:

1. Do first generation OTC antihistamines make voice function worse as measured via voice acoustic and aerodynamic measures? It is hypothesized that all objectives measures will reflect a negative change in voice function.
2. Do first generation OTC antihistamines make voice function worse as measured via participant and researcher perceptual measures? It is hypothesized that participants will rate their vocal function as more effortful after taking the antihistamine and researchers will rate voice quality as worse.

Participants ages 18-35 who have been diagnosed with allergies, are free of laryngeal pathology, and meet inclusion criteria will be consented. Participation in the study involves a pretrial visit and one day of data collection. The initial visit will obtain informed consent and train the trial measures. The 2nd day involves determination of systemic hydration (<1.02 g/ml), administration of the OTC antihistamine (Chlor-Trimeton), and measures taken at baseline and 3 hours after antihistamine administration. This antihistamine was selected for its lower sedation and anticholinergic effects than its other first-generation options. Each participant will take one, 12mg tablet. Onset action time for this antihistamine is 3 hours. Participants will be given water to consume during the 3 hour wait for the 2nd data time point to maintain hydration. Measures include routine clinical perceptual, acoustic, aerodynamic, and laryngeal imaging measures.

DETAILED DESCRIPTION:
Using a within-participant repeated measures design, ten 18-35-year-old males and females will be recruited locally to participate in this preliminary study. This age range was selected to assure laryngeal maturity following adolescence and avoid musculoskeletal/hormonal changes secondary to perimenopause. Informed consent will be obtained from each participant prior to screening for eligibility. Inclusion criteria: the ability to match pitch on a screening task, have diagnosed allergies of the upper airway, a Sino-nasal Outcome Test( SNOT-22) score of 20 or greater, pass videostroboscopic prescreening for laryngeal pathologies, no history of voice disorder, ability to comfortably breathe through both their nose and mouth, no history of drying medications other than the antihistamine, reflux, respiratory diseases, diabetes, neurological problems, hormone imbalance, pregnancy, breastfeeding over the preceding 6 months, or active smoker at the time of investigation. Participation in the study involves a pretrial visit and one day of data collection.

At the pretrial visit the participants will be screened for fever, cough, and other flu like symptoms using the screening questions outlined via Auburn's Human Research COVID-19 matrix. If a participant answers "yes" to any of the questions, the pretrial visit will be cancelled or postponed to a later day.

The pre-trial training visit will take place in the Auburn University Department of Speech, Language, and Hearing Sciences Voice Physiology Laboratory. If the participant passes the screener the pre-trial visit will include 1) the informed consent process, 2) collection of demographic data (age, sex, racial and ethnic identity, medications, time of day for medication intake), 3) the participant completing the SNOT-22, 4) completion of a routine laryngeal and vocal fold screening, and 5) training for the routine clinical acoustic and aerodynamic tasks. The laryngeal screening will be done by a trained speech-language pathologist in accordance with standard and routine laryngeal imaging procedures. Volunteers will be asked if they are allergic to topical Hurricaine spray. Volunteers unable to tolerate the procedure without application of topical anesthetic Hurricaine spray or allergic to Hurricaine spray will be thanked for their interest and dismissed from the study. Volunteers showing evidence of laryngeal pathology will be dismissed from the investigation and referred to their primary care provider.

The day prior to the trial visit the participants will be screened remotely via phone for fever, cough, and other flu like symptoms using the screening questions outlined via Auburn's Human Research COVID-19 matrix. If a participant answers "yes" to any of the questions, the trial visit will be cancelled and postponed to a later day. Participants will be reminded to wear a mask and/or face covering should that be required via application of the Auburn University COVID-19 matrix.

The trial visit will occur in Auburn University Speech and Hearing Clinic in the Voice Physiology Lab. Trial visits will be completed close to the same time of day across all participants to avoid variables associated with circadian rhythm.

1. A urine sample will be obtained for specific gravity analysis, a routine objective measurement of systemic hydration, via reagent strip for urinalysis (Siemens Multistix® 10 Specific Gravity Urine Test Strips, USA). A value of ≤ 1.020g/ml is a well-established threshold of appropriate systematic hydration. It is critical that adequate systemic hydration be established to ensure that the research variables of interest are due to the antihistamine drying effects. If a participant is not adequately hydrated, they will be asked to drink water until hydration criterion is achieved.
2. Participants will then complete a routine laryngeal and vocal fold screening. The laryngeal screening will be done in accordance with standard and routine laryngeal imaging procedures and will be completed by a speech-language pathologist who routinely conducts this procedure.
3. Participants will then complete the OMNI-Vocal Effort Scale (OMNI-VES) and the Rating-of-Fatigue Scale (ROF).
4. Acoustic parameters will then be collected using routine clinical measures within PRAAT (version 6.1.03), using a headset microphone placed 2 cm from the corner of the mouth. The participant will read standard sentences at conversational pitch and loudness and the following measures will be derived: speaking fundamental frequency and cepstral peak prominence (CPP). The participant will also be asked to sustain the vowel "a" at normal pitch and conversational loudness to determine the following: harmonic to noise ratio and mean fundamental frequency. All acoustic files will be saved under participant number and saved on a password protected share drive.
5. Aerodynamic measures will be collected using the PENTAX Phonatory Aerodynamic System (PAS) to assess phonation threshold pressure (PTP) using well-established standard routine clinical procedures. Aerodynamic measures are collected with a face mask and oral pressure tube that collect airflow and air pressure for a standard task.

After collecting the baseline measures for the participant, they will be administered the first-generation antihistamine, Chlor-Trimeton, at the recommended packaging dose, one, 12mg tablet. The onset of action time, the length of time it takes for the medication to start to work, for this antihistamine is 3 hours. During the 3 hours, the participant will be asked to sit and remain as quiet as possible. The participant is free to study or quietly use electronic during this period. The participant will also be instructed to drink a bottle of water to maintain their baseline hydration based on their age and sex. After the 3 hour time period has concluded, all perceptual, acoustic, aerodynamic, and laryngeal imaging measures will be completed again. This trial visit will take 4 hours. Total participant time will be approximately 5 hours for this study.

ELIGIBILITY:
Inclusion Criteria:

* the ability to match pitch on a screening task
* have diagnosed allergies of the upper airway
* a SNOT-22 score of 20 or greater (19)
* pass videostroboscopic prescreening for laryngeal pathologies
* no history of voice disorder
* ability to comfortably breathe through both their nose and mouth
* no history of drying medications other than the antihistamine, reflux, respiratory diseases, diabetes, neurological problems, hormone imbalance, pregnancy, breastfeeding over the preceding 6 months, or active smoker at the time of investigation.

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Urine specific gravity (g/ml) | Start of trial
  Objective measurement of systemic hydration
Fundamental frequency (Hertz) | Change from Baseline Fundamental Frequency at 3 hours
  Sustained "a" task from which the cycles of vocal fold vibration per second are extracted.
Speaking fundamental frequency (Hertz) | Change from Baseline Fundamental Frequency at 3 hours
  Standard reading task from which the average cycles per second of vocal fold vibration are extracted.
Harmonic-to-Noise ratio (decibels, dB) | Change from Baseline Fundamental Frequency at 3 hours
  Sustained "a" task from which a ratio of the harmonic acoustic components of the signal relative to the noise components of the acoustic signal are determined
Cepstral peak prominence (decibels, dB) | Change from Baseline Fundamental Frequency at 3 hours
  An acoustic measurement of voice quality deviation that is extracted from a recorded speech sample.
Phonation threshold pressure (cm/H20) | Change from Baseline Fundamental Frequency at 3 hours
  An aerodynamic measurement of the minimum amount of subglottal pressure required to initiate vocal fold vibration for voicing
Videostroboscopy (video of vocal fold vibration) | Change from Baseline Fundamental Frequency at 3 hours
  Standard clinical endoscopic imaging of laryngeal structure and function
OMNI-Vocal Effort Scale (scaled score) | Change from Baseline Fundamental Frequency at 3 hours
  A validated scale of perceived vocal effort that provides a scale of 1-10 from which to determine how much vocal effort was produced.
Rating-of-Fatigue (ROF; scaled score) | Change from Baseline Fundamental Frequency at 3 hours
  A validated scale of perceived voice fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Sandage, PhD, Principal Investigator — Auburn University
Locations (1):
- Department of Speech, Language & Hearing Sciences, Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No